CLINICAL TRIAL: NCT05473455
Title: Does Addition of Follicular Flushing to the Initial Aspiration Lead to Higher Numbers of Oocytes Retrieved in Women Undergoing Oocyte Retrieval? A Randomized Controlled Trial
Brief Title: Value of Follicular Flushing. Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Flushing RCT
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Infertility
Keywords: Follicular Flushing; Oocyte Retrieval
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follicular aspiration with addition of follicular flushing. (Experimental): All follicles will be aspirated with the addition of follicular flushing if necessary (up to 5 times per follicle)
  Interventions: Procedure: Experimental: Follicular aspiration with addition of follicular flushing.
- Follicular aspiration only. (No Intervention): All follicles will be aspirated and no flushing will be applied.

INTERVENTIONS:
Procedure: Experimental: Follicular aspiration with addition of follicular flushing. — Follicular flushing if necessary up to 5 times using a double lumen needle for oocyte recovery
  Arms: Follicular aspiration with addition of follicular flushing.

SUMMARY:
The purpose of this study is to evaluate whether the addition of follicular flushing to the initial aspiration during oocyte retrieval increases the number of oocytes retrieved in women undergoing ovarian stimulation.

DETAILED DESCRIPTION:
There is an ongoing debate regarding the effectiveness of follicular flushing during oocyte retrieval. Currently published studies and metanalyses suggest that follicular flushing does not improve live birth rate, clinical pregnancy rate or the number of oocytes retrieved. However, currently published studies may be confounded by the types of needle used, aspiration pressures, number of times flushing is repeated, etc. Additionally, follicular flushing should be examined in specific patient populations according to their response to ovarian stimulation.

In the current study, each woman will have one ovary (right or left) randomly assigned to be aspirated with or without the addition of follicular flushing. This study design ensures that clinical and demographic characteristics of the couple will not affect the outcomes evaluated. The primary endpoints will be the number of oocytes retrieved per ovary assigned to each group. Secondary outcomes will be the oocyte recovery rate (oocytes retrieved per follicle aspirated) oocyte maturation rate, fertilization rate, and embryo development per ovary assigned to each group.

The study population will include three subgroups according to observed ovarian response to ovarian stimulation (poor responders, normal responders, hyper responders). Assuming a minimum clinically significant difference in oocyte yield of 1 oocyte, a sample size of twenty patients per subgroup is required to yield 80% power.

Patients aged <43 years with the presence of at least one follicles >11mm in each ovary on the day of triggering final oocyte maturation will be eligible for inclusion in the study. 60 patients (20 in each of the aforementioned subgroup) will be recruited and just prior to oocyte retrieval their left and right ovaries will be randomly allocated into flushing or the no-flushing group. In both ovaries all follicles greater than 11mm will be punctured by the same 16G double lumen needle, using the same aspiration pressure. In the flushing group, flushing will be performed up to a maximum of five times or until a cumulus oocyte complex (COC) is retrieved.

In the control group all follicles greater than 11mm will be aspirated by the same double lumen needle and no flushing will be performed.

All COCs will be grouped according to the ovary they originated from by the embryologists and their development will be recorded until Day 3 following fertilization (Number of MII oocytes, number of fertilized oocytes, number good quality Day 3 embryos).

ELIGIBILITY:
Inclusion Criteria:

* Presence of both ovaries
* 18-43 years old
* At least one follicle >11mm present in each ovary on day of triggering final oocyte maturation.

Exclusion Criteria:

* Ovarian surgery
* Monofolicular development

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants must have both ovaries present
Enrollment: 105 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | During oocyte collection (usually 10-30 minutes)
  Number of oocytes retrieved per ovary randomised

SECONDARY OUTCOMES:
Oocyte recovery rate | During oocyte collection (usually 10-30 minutes)
  Number of oocytes retrieved per follicle aspirated
Oocyte maturation rate | During oocyte denudation (usually 10-30 minutes)
  Number of mature (metaphase-II) oocytes divided by the number of oocytes retrieved per ovary randomised
Fertilization rate | During fertilisation check (usually 10 minutes)
  Number of fertilised (2PN) oocytes divided by the number of matured oocytes retrieved per ovary randomised
Percentage of good quality embryos on day 2/3 | During embryo evaluation (usually 10 minutes)
  Number of good quality embryos divided by the number of fertilized oocytes per ovary randomised

CONTACTS AND LOCATIONS:
Overall Officials: Lainas, PhD, Study Director — Eugonia
Locations (1):
- Eugonia Unit of Assisted Reproduction, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Horn K, Depenbusch M, Schultze-Mosgau A, Griesinger G. Randomized, open trial comparing a modified double-lumen needle follicular flushing system with a single-lumen aspiration needle in IVF patients with poor ovarian response. Hum Reprod. 2017 Apr 1;32(4):832-835. doi: 10.1093/humrep/dex019. PMID 28333185
- [Background] Franasiak JM. Follicular flushing: time to look elsewhere to improve in vitro fertilisation outcomes? BJOG. 2017 Jul;124(8):1197. doi: 10.1111/1471-0528.14628. No abstract available. PMID 28276189
- [Background] Roque M, Sampaio M, Geber S. Follicular flushing during oocyte retrieval: a systematic review and meta-analysis. J Assist Reprod Genet. 2012 Nov;29(11):1249-54. doi: 10.1007/s10815-012-9869-9. Epub 2012 Oct 13. PMID 23065177
- [Derived] Lainas GT, Lainas TG, Makris AA, Xenariou MV, Petsas GK, Kolibianakis EM. Follicular flushing increases the number of oocytes retrieved: a randomized controlled trial. Hum Reprod. 2023 Oct 3;38(10):1927-1937. doi: 10.1093/humrep/dead169. PMID 37632249